CLINICAL TRIAL: NCT07036055
Title: Targeting Brain-Heart Coupling to Improve Emotional Inhibitory Control in Alcohol Use Disorder: Mechanistic Insights and Effects of Transcutaneous Auricular Vagus Nerve Stimulation Combined With Mindfulness Training
Brief Title: Research on the Heart-Brain Coupling Mechanisms and Interventions for Emotional Inhibitory Control Deficits in Individuals With Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JDu-015
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorder (AUD); transcutaneous auricular vagus nerve stimulation (taVNS); brain-heart coupling; mindfulness meditation
MeSH Terms: conditions — Alcoholism | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS + Mindfulness Training (Experimental): Participants in this group will receive 30-minute daily sessions of transcutaneous auricular vagus nerve stimulation (taVNS) combined with standardized mindfulness training for 10 consecutive days. taVNS is delivered using a wearable device targeting the cymba conchae area of the ear. Stimulation parameters include a frequency of 25 Hz and a pulse width of 200 µs. Mindfulness training involves guided audio practice focused on breath awareness and body scanning.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS); Behavioral: Mindfulness Training
- Sham Stimulation + Mindfulness Training (Sham Comparator): Participants in this group will receive 30-minute daily sessions of sham stimulation (identical device without active current) combined with the same mindfulness training protocol as the experimental group, administered for 10 consecutive days. The sham stimulation mimics the appearance and procedure of active taVNS but delivers no electrical stimulation.
  Interventions: Device: Sham Stimulation; Behavioral: Mindfulness Training

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — Participants receive transcutaneous auricular vagus nerve stimulation (taVNS) via a non-invasive ear-clip device targeting the cymba conchae. The device delivers electrical pulses at 25 Hz frequency with a pulse width of 200 µs, for 30 minutes daily over 10 consecutive days. The stimulation intensity is individually adjusted to the participant's perceptual threshold. taVNS is paired with standardized mindfulness training in this arm.
  Other Names: taVNS; Auricular Vagus Nerve Stimulation
  Arms: taVNS + Mindfulness Training
Device: Sham Stimulation — Participants in this group use the same device as in the active taVNS condition, but the stimulation is deactivated. The ear-clip device is placed identically on the cymba conchae, with no electrical current delivered. This sham procedure mimics the look and feel of taVNS but serves as a placebo control. Sham stimulation is combined with the same mindfulness training as the experimental group.
  Arms: Sham Stimulation + Mindfulness Training
Behavioral: Mindfulness Training — Participants receive instructor-led mindfulness training conducted by a trained therapist. Each session lasts 30 minutes and focuses on breath awareness, body scanning, and non-judgmental awareness of internal experience. All participants (both taVNS and sham groups) receive this training daily for 10 consecutive days.
  Other Names: Mindfulness Meditation; Guided Mindfulness Practice

SUMMARY:
The goal of this clinical trial is to understand whether combining transcutaneous auricular vagus nerve stimulation (taVNS) with mindfulness training can improve emotional inhibitory control in adults with Alcohol Use Disorder (AUD). The study also aims to explore the brain-heart coupling mechanisms underlying these control deficits.

The main questions it aims to answer are:

Do individuals with AUD have abnormal brain-heart coupling associated with impaired emotional inhibitory control? Can taVNS combined with mindfulness training enhance emotional inhibitory control in individuals with AUD compared to sham stimulation? Researchers will compare a group receiving taVNS plus mindfulness training to a group receiving sham stimulation plus mindfulness training to see whether the active intervention improves behavioral performance and brain-heart coupling.

Participants will:

Complete an emotional Go/NoGo task while EEG and ECG data are recorded Receive 10 days of either real or sham taVNS combined with mindfulness training Complete questionnaires and cognitive assessments before and after the intervention

DETAILED DESCRIPTION:
This two-part clinical study investigates the mechanisms and intervention effects related to emotional inhibitory control deficits in individuals with Alcohol Use Disorder (AUD), with a specific focus on brain-heart coupling (also referred to as brain-heart interplay, BHI). The study aims to identify the neurophysiological characteristics underlying inhibitory control impairments in AUD and evaluate whether non-invasive vagus nerve stimulation combined with mindfulness training can enhance emotional regulation and cognitive function.

Study 1: Mechanism Exploration Study 1 adopts a case-control observational design. A total of 28 individuals diagnosed with AUD (based on DSM-5 criteria) and 28 age- and education-matched healthy controls are recruited. Participants complete an emotional Go/NoGo task under EEG-ECG hyperscanning. Emotional inhibitory control performance is assessed through behavioral indices (reaction time, error rate) and further analyzed using the Hierarchical Drift Diffusion Model (HDDM) to quantify latent cognitive processing parameters (e.g., drift rate, boundary separation, non-decision time). Brain-heart coupling is evaluated through resting-state EEG-ECG data using multiscale coupling coefficients and maximal information coefficient (MIC) between heart rate variability (HRV) and cortical oscillations (particularly α, β, and θ bands).

Primary outcomes include:

Drift rate and inhibitory control accuracy under emotional interference Degree of BHI (HRV-EEG coupling strength and directionality) The moderating effect of self-reported emotion regulation ability (measured via DERS)

Study 2: Intervention Evaluation

Study 2 is a single-blind randomized controlled trial (RCT) involving 60 AUD participants randomly assigned to:

Active group (n=30): taVNS combined with mindfulness training Control group (n=30): sham stimulation combined with mindfulness training Participants in both groups receive daily 30-minute sessions for 10 consecutive days. taVNS is delivered using a wearable ear-clip device targeting the auricular branch of the vagus nerve (cymba conchae), with stimulation parameters set at 25 Hz, pulse width of 200 μs, and intensity adjusted to individual sensory threshold. Mindfulness training is conducted by a trained therapist, focusing on breath awareness and body scanning.

Outcome measures are collected pre- and post-intervention and include:

Emotional inhibitory control performance under the Go/NoGo paradigm HDDM-derived cognitive parameters (e.g., drift rate) EEG-ECG-based BHI metrics (HRV-EEG coupling during rest) Self-reported anxiety (GAD-7), depressive symptoms (PHQ-9), and alcohol craving Adverse events monitoring and adherence logs Data Acquisition and Processing EEG signals are recorded using a 64-channel portable system (10-20 system); ECG is simultaneously recorded.

Signals are preprocessed in EEGLAB (bandpass filtering, artifact correction via ASR), with HRV features extracted via Kubios.

HDDM modeling is conducted in Python (Bayesian MCMC estimation), and BHI is analyzed through mutual information, MIC, and transfer entropy metrics.

Sample Size and Statistical Plan Sample size was estimated based on prior effect sizes observed in similar taVNS and mindfulness interventions. Power analysis indicated 28 subjects per group achieves >80% power to detect moderate group × time interaction effects.

Statistical analyses include:

Mixed-effects ANOVA for behavioral and neural outcomes Regression models to assess mediation and moderation effects (e.g., emotion regulation ability) Pearson/Spearman correlation between physiological and behavioral measures All analyses follow intention-to-treat principles with imputation for missing data where appropriate (e.g., multiple imputation for <10% missing).

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-5 diagnostic criteria for Alcohol Use Disorder (AUD).
2. Aged 18-55 years.
3. Currently in the post-acute withdrawal phase (≥2 weeks since last alcohol use).
4. No severe psychiatric comorbidities (e.g., schizophrenia, bipolar disorder).
5. No neurological disorders (e.g., epilepsy, traumatic brain injury).
6. Willing to provide informed consent.

Exclusion Criteria:

1. Dependence on other substances (except nicotine).
2. Severe physical illness requiring immediate treatment.
3. Active infectious diseases (e.g., HIV, hepatitis).
4. Inability to complete study procedures (e.g., cognitive impairment).

*(For healthy controls in Study 1, inclusion required AUDIT score ≤8, no psychiatric/neurological history, and matched demographics.)*

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Emotional Inhibitory Control Performance in Emotional Go/NoGo Task | Assessed at baseline (Day 0) and post-intervention (Day 11)
  Emotional inhibitory control performance will be assessed based on participants' accuracy in the emotional Go/NoGo task (i.e., proportion of correctly inhibited responses on NoGo trials). The task uses emotionally valenced facial stimuli and requires participants to withhold responses under emotional interference. Accuracy reflects participants' inhibitory control under affective load, which is the primary behavioral index of intervention efficacy.

SECONDARY OUTCOMES:
Drift Rate Estimated by Hierarchical Drift Diffusion Model (HDDM) | Assessed at baseline (Day 0) and post-intervention (Day 11)
  Drift rate, a latent parameter derived from the HDDM, reflects the efficiency of cognitive processing and evidence accumulation during the Go/NoGo task. Higher drift rate indicates more efficient response selection under emotional conflict. HDDM modeling is conducted using trial-level reaction time and accuracy data.
Brain-Heart Coupling Strength (HRV-EEG Coupling) | Assessed at baseline (Day 0) and post-intervention (Day 11)
  Degree of brain-heart coupling is measured by calculating multiscale mutual information and maximal information coefficient (MIC) between heart rate variability (HRV) and EEG oscillations (particularly in the alpha, beta, and theta bands) during resting-state data collection. Higher coupling indicates stronger brain-autonomic integration.
Self-Reported Emotion Regulation Ability (DERS Score) | Assessed at baseline (Day 0) and post-intervention (Day 11)
  Participants complete the Difficulties in Emotion Regulation Scale (DERS), which provides a total score and subscale scores reflecting emotional awareness, impulse control, and clarity. Lower scores reflect better emotion regulation capacity.
Alcohol Craving (Visual Analog Scale) | Assessed at Day 0, Day 3, Day 6, Day 11
  Alcohol craving is measured using a visual analog scale (VAS, 0-100), with higher scores indicating stronger desire to consume alcohol. This outcome reflects emotional-behavioral change after intervention.

OTHER OUTCOMES:
Anxiety Symptoms (GAD-7 Score) | Assessed at Day 0, Day 3, Day 6, Day 11
  Participants complete the Generalized Anxiety Disorder 7-item scale (GAD-7). Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Depressive Symptoms (PHQ-9 Score) | Assessed at Day 0, Day 3, Day 6, Day 11
  Participants complete the 9-item Patient Health Questionnaire (PHQ-9). Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D, Study Chair — Shanghai Mental Health Center
Locations (1):
- China, Mengzi, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the published results, including behavioral performance, physiological signals (EEG/ECG), and questionnaire scores, will be shared in de-identified form. Data dictionaries will also be provided.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be available starting 6 months after publication of the primary results and will remain available for 3 years.
Access Criteria: IPD will be shared with qualified researchers affiliated with academic or non-profit institutions, for secondary analyses that are methodologically sound and ethically approved. Requests will be reviewed by the principal investigator and must include a study proposal, data use agreement, and proof of institutional ethics approval.